CLINICAL TRIAL: NCT00849550
Title: A Phase I Study of Capecitabine, Oxaliplatin, Bevacizumab, and RAD001 (XELOX-A-Ev) for Subjects With Advanced Solid Tumors
Brief Title: Safety and Dosage Study of RAD001 (Everolimus) in Combination With Current Standard of Care to Treat Advanced Solid Tumors.
Acronym: COBRA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Herbert Hurwitz (Other)
Collaborators: Roche-Genentech (Industry); Novartis (Industry)
Responsible Party: Sponsor-Investigator, Herbert Hurwitz, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00015605; 4265 (Other: Legacy IRB number)
Record Dates: First submitted 2009-02-22; First posted 2009-02-24 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific; Cancer
Keywords: Advanced Solid Tumors; Cancer; Capecitabine; XELOX; Neoplasms; Oxaliplatin; Bevacizumab; RAD001
MeSH Terms: conditions — Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- XELOX-A-Ev (Experimental)
  Interventions: Drug: capecitabine/oxaliplatin/bevacizumab/RAD001 (XELOX-A-Ev)

INTERVENTIONS:
Drug: capecitabine/oxaliplatin/bevacizumab/RAD001 (XELOX-A-Ev) — bevacizumab IV, capecitabine oral, oxaliplatin IV, RAD001 oral

SUMMARY:
The purpose of this study is to determine if RAD001 (everolimus) helps improve the standard treatment of XELOX-A (bevacizumab, oxaliplatin, capecitabine) in advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years or older
* Must have a performance status of at least 70% (able to carry on most normal activities)
* Must have life expectancy of at least 3 months
* Must have adequate organ and marrow function as determined by lab tests
* Women of child-bearing potential and men must agree to use two forms of contraception
* Ability and willingness to sign a written informed consent document
* Histologically confirmed solid tumor malignancy that is metastatic or unresectable

Exclusion Criteria:

* Pregnant or breastfeeding and/or lactating women
* Patients who have received any other investigational agents within 28 days of the first day of study drug
* Patients with known CNS metastases
* History of other carcinomas within last 5 years (except non-melanoma skin cancer, in-situ cervical cancer, localized prostate cancer)
* Inadequately controlled hypertension
* Significant vascular disease
* Invasion or encasement of a major artery
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to day 1 of study drug
* Serious illness or medical condition
* History of myocardial infarction, unstable angina, cardiac or other vascular stenting
* History of stroke
* HIV, Hepatitis C, Hepatitis B or other serious chronic infection
* Impairment of Gastrointestinal function or disease
* History of interstitial lung disease
* Patients who have had radiation therapy, hormonal therapy, biologic therapy or chemotherapy for cancer within 28 days of receiving study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To determine the MTD/RPTD of capecitabine/oxaliplatin/bevacizumab/everolimus (XELOX-A-Ev) for subjects with advanced solid tumors. | End of treatment phase

SECONDARY OUTCOMES:
Describe dose-limiting and non-dose-limiting toxicities | End of treatment phase
preliminarily investigate the response rate and PFS | from response to progression

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Hurwitz, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Ingalls Cancer Research Center, Harvey, Illinois
  - Duke University Medical Center, Durham, North Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee